CLINICAL TRIAL: NCT03287440
Title: Pilot Study of Rehabilitation in Safety-net Settings for Patients With COPD
Brief Title: Rehabilitation for Patients With COPD
Acronym: COPD Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other); Nina Ireland Program in Lung Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Health Services Research
Other Study IDs: 16-19967
Record Dates: First submitted 2017-09-05; First posted 2017-09-19 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Health Disparities; Lung Diseases; Self-management; Chronic Disease; Socio-economic status
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Chronic Disease

STUDY DESIGN:
Intervention Model Description: A step-wedge design will allow all participants to receive the intervention. Participants not immediately enrolled into the intervention will serve as controls. At the time of the intervention, these participants will move over to the treatment arm.
  The first two groups will be used to refine the COPD Wellness intervention and identify social barriers specific to individuals living with COPD. Starting with group 3, we will alternate the addition of the Health Advocates (HA) program as an adherence strategy in order to determine the HA's effect on participation in COPD Wellness.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator and outcome assessor will be masked to when the participant completes the intervention and to whether or not they received the Health Advocates adherence strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD Wellness With Health Advocate (Active Comparator): This arm will be given low-intensity pulmonary rehabilitation, COPD Wellness, for individuals with moderate-to-severe COPD with an additional assignment of a health advocate to address unmet social needs as an adherence strategy.
  Interventions: Behavioral: COPD Wellness; Behavioral: Health Advocate
- COPD Wellness (Active Comparator): This arm will only be given low-intensity pulmonary rehabilitation, COPD Wellness, for individuals with moderate-to-severe COPD.
  Interventions: Behavioral: COPD Wellness

INTERVENTIONS:
Behavioral: COPD Wellness — This is low-intensity pulmonary rehabilitation that incorporates exercise, nutrition, patient education, and a support group class.
Behavioral: Health Advocate — The Zuckerberg San Francisco General (ZSFG) Hospital Health Advocates program links social needs screening with a tiered referral and linkage process to appropriate resources
  Arms: COPD Wellness With Health Advocate

SUMMARY:
This study will examine COPD Wellness, a 10-week low-intensity pulmonary rehabilitation program consisting of group and home exercise, education, and social support can improve symptoms and increase physical activity in participants with COPD who receive care within a 'safety-net' healthcare system (e.g. County Hospital). Half of the participants will also receive an adherence strategy targeted at addressing unmet social needs, while the other half will undergo the intervention without the adherence strategy.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD), one of the leading causes of death in the US, disproportionately affects low socioeconomic communities. While few interventions effectively modify the course of COPD and improve outcomes, pulmonary rehabilitation is the one notable exception. However, implementation of this resource-intensive program in real-life settings, and in particular, for underserved communities, has proven to be challenging. Safety-net centers that serve primarily under-insured populations lack financial resources to provide pulmonary rehabilitation.

COPD Wellness, a 10-week low-intensity pulmonary rehabilitation program consisting of group and home exercise, education, and social support, was developed to address this gap. This intervention is targeted at patients with moderate to severe COPD (GOLD Class B-D) who receive care through a safety-net health system. To be impactful, risk factors for low adherence include both disease severity and socio-environmental factors, must be addressed. As merely having a pulmonary rehabilitation program will not automatically lead to improved outcomes.

As part of this study, an adherence strategy targeted at addressing unmet social needs to improve health will also be implemented. A Health Advocates program that links social needs screening with a tiered referral and linkage process to appropriate resources will be tested to see if adherence to COPD Wellness (exercise intervention) improves by addressing competing non-medical stressors.

ELIGIBILITY:
Inclusion Criteria:

* Age: Are greater than or equal to 40 years
* Diagnosis: COPD Gold Stage Class B-D (symptomatic disease), COPD/Asthma overlap with symptoms
* Language: English
* Care Center: ZSFG, Community Health Center clinics, Federally Qualified Health Centers
* Availability: Able to participate in a 10-week, weekly course at the weekly scheduled time (can defer x 1)

Exclusion Criteria:

* Planning to move out of the area within the next year
* Eligible for and desire to go to full intensity pulmonary rehabilitation. Participant has Medicare Part A and B OR have San Francisco Health Plan. For those that met these criteria, we will assist with referral to program
* Resides in any kind of long-term care facilities that is NOT Laguna Honda or the Mental Health Rehabilitation Facility
* Has a diagnosis of interstitial lung disease, pulmonary fibrosis, or cystic fibrosis
* Active, chronic lung infection, such as tuberculosis
* A history of a pulmonary embolism in the year (12 months) prior to recruitment
* History of a myocardial infarction in the year (12 months) prior to recruitment
* In the 12 weeks prior to recruitment, has had history of unstable heart disease (including valve disease), heart failure, or uncontrolled irregular heart beat

Potential participants who have had the following will be re-assess for eligibility 6 weeks after the initial assessment:

* A pulmonary exacerbation or worsening of COPD/Asthma symptoms in the past 6 weeks
* History of an upper respiratory infection in the past 6 weeks
* History of an eye, chest, or abdominal surgery within the past 6 weeks

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline 6 Minute Walk Test at End of Intervention | End of Intervention, an average of 4 months
  Standardized test to measure distance walked in 6 minutes
Change from Baseline COPD Assessment Test (CAT) at End of Intervention | End of Intervention, an average of 4 months
  Questionnaire assessing COPD symptoms and quality of life

SECONDARY OUTCOMES:
Change from Baseline number of exacerbations of COPD at End of Intervention | End of Intervention, an average of 4 months
  Exacerbation defined as a visit to an urgent care or emergency department for COPD, a hospitalization for COPD, or a prescription of an oral steroid for worsening COPD symptoms
Change from Baseline number of exacerbations of COPD at 12 months | 12 months
  Exacerbation defined as a visit to an urgent care or emergency department for COPD, a hospitalization for COPD, or a prescription of an oral steroid for worsening COPD symptoms
Change in baseline Smoking status at end of intervention | End of Intervention, an average of 4 months
  Have you smoked a cigarette in the past 30 days
Change in baseline Smoking status at 12 months | 12 months
  Have you smoked a cigarette in the past 30 days
Change from baseline D-12 evaluation at end of intervention | End of Intervention, an average of 4 months
  Evaluates dyspnea symptoms and increased ease of activities of daily living as related to COPD symptoms
Change from baseline D-12 evaluation at 12 months | 12 months
  Evaluates dyspnea symptoms and increased ease of activities of daily living as related to COPD symptoms
Change in baseline Patient Health Questionnaire (PHQ-)8 at End of Intervention | End of Intervention, an average of 4 months
  Diagnoses of depressive disorders and depression severity
Adherence | Assessed during 10-week COPD Wellness Intervention
  Number of classes attended by the participant
Change from Baseline 6 Minute Walk Test at 12 months | Baseline and 12 months
  Standardized test to measure distance walked in 6 minutes
Change from Baseline COPD Assessment Test (CAT) at 12 months | Baseline, 12 months
  Measure of COPD symptoms and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Thakur, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Troosters T, Gosselink R, Decramer M. Short- and long-term effects of outpatient rehabilitation in patients with chronic obstructive pulmonary disease: a randomized trial. Am J Med. 2000 Aug 15;109(3):207-12. doi: 10.1016/s0002-9343(00)00472-1. PMID 10974183
- [Background] Baumann HJ, Kluge S, Rummel K, Klose H, Hennigs JK, Schmoller T, Meyer A. Low intensity, long-term outpatient rehabilitation in COPD: a randomised controlled trial. Respir Res. 2012 Sep 27;13(1):86. doi: 10.1186/1465-9921-13-86. PMID 23017153
- [Background] Selzler AM, Simmonds L, Rodgers WM, Wong EY, Stickland MK. Pulmonary rehabilitation in chronic obstructive pulmonary disease: predictors of program completion and success. COPD. 2012 Aug;9(5):538-45. doi: 10.3109/15412555.2012.705365. PMID 23030585
- [Background] Fischer MJ, Scharloo M, Abbink JJ, van 't Hul AJ, van Ranst D, Rudolphus A, Weinman J, Rabe KF, Kaptein AA. Drop-out and attendance in pulmonary rehabilitation: the role of clinical and psychosocial variables. Respir Med. 2009 Oct;103(10):1564-71. doi: 10.1016/j.rmed.2008.11.020. Epub 2009 May 29. PMID 19481919
- [Background] Rochester CL, Vogiatzis I, Holland AE, Lareau SC, Marciniuk DD, Puhan MA, Spruit MA, Masefield S, Casaburi R, Clini EM, Crouch R, Garcia-Aymerich J, Garvey C, Goldstein RS, Hill K, Morgan M, Nici L, Pitta F, Ries AL, Singh SJ, Troosters T, Wijkstra PJ, Yawn BP, ZuWallack RL; ATS/ERS Task Force on Policy in Pulmonary Rehabilitation. An Official American Thoracic Society/European Respiratory Society Policy Statement: Enhancing Implementation, Use, and Delivery of Pulmonary Rehabilitation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1373-86. doi: 10.1164/rccm.201510-1966ST. PMID 26623686